CLINICAL TRIAL: NCT03180216
Title: Novel Antigens Targeted by Ex Vivo Expanded T-Lymphocytes for Prevention or Treatment of Viral Infections Following Hematopoietic Stem Cell Transplantation
Brief Title: T-Lymphocytes for Prevention or Treatment of Viral Infections Following Hematopoietic Stem Cell Transplantation
Acronym: NATS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Michael Keller, Assistant Professor, Division of Allergy / Immunology, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008637
Record Dates: First submitted 2017-05-01; First posted 2017-06-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Viral Infections; Bone Marrow Transplant Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prophylactic and treatment (Experimental): Virus Specific T cells (VSTs) for prophylactic and treatment of active viral infection(s) after HSCT.
  3 different dose levels starting with 1 x 10E7 /m2 (a T cell number more than an order of magnitude lower than that administered at the time of an unmanipulated marrow infusion), followed by 2 x 10E7/m2 and a final dose 5 x 10E7 VSTs/m2
  Interventions: Biological: Virus Specific T cells (VSTs)

INTERVENTIONS:
Biological: Virus Specific T cells (VSTs) — This Phase I dose-escalation trial is designed to evaluate the safety of rapidly generated multivirus-specific T-cell products with antiviral activity against CMV, EBV, adenovirus, HHV6, BK virus, JC virus, and human parainfluenza-3 (HPIV3), derived from eligible HSCT donors.
  In this trial, we will utilize a rapid generation protocol for broad spectrum multivirus-specific T cells for infusion to recipients of allogeneic hematopoietic stem cell transplant (HSCT), who are at risk of developing EBV, CMV, adenovirus, HHV6, BKV, JCV and/or HPIV3, or with PCR/culture confirmed active infection(s) of EBV, CMV, adenovirus, HHV6, BKV, JCV, and/or HPIV3 that has failed to resolve with at least 14 days of standard antiviral therapy (if available and tolerated). These cells will be derived from HSCT donors, and the study agent will be assessed at each dose for evidence of dose-limiting toxicities (DLT).

SUMMARY:
This Phase I dose-escalation trial is designed to evaluate the safety of rapidly generated multivirus-specific T-cell products with antiviral activity against CMV, EBV, adenovirus, HHV6, BK virus, JC virus, and human parainfluenza-3 (HPIV3), derived from eligible HSCT donors.

In this trial, we will utilize a rapid generation protocol for broad spectrum multivirus-specific T cells for infusion to recipients of allogeneic hematopoietic stem cell transplant (HSCT), who are at risk of developing EBV, CMV, adenovirus, HHV6, BKV, JCV and/or HPIV3, or with PCR/culture confirmed active infection(s) of EBV, CMV, adenovirus, HHV6, BKV, JCV, and/or HPIV3 that has failed to resolve with at least 14 days of standard antiviral therapy (if available and tolerated). These cells will be derived from HSCT donors, and the study agent will be assessed at each dose for evidence of dose-limiting toxicities (DLT).

This study will have two arms: Arm A will include patients who receive prophylactic treatment, and Arm B will include patients who receive VSTs for one or more active infections with targeted viruses. Determination of the study arm will be determined by the patient's clinical status. Study arms will each be analyzed for safety endpoints and secondary endpoints.

DETAILED DESCRIPTION:
Viral infections are normally controlled by T-cell immunity and are a cause of significant morbidity and mortality during the period of immune recovery after hematopoietic stem cell transplantation (HSCT). Risk for infection is impacted by the degree of tissue mismatch between donor and recipient and the immune status of the donor, including the degree and length of immunosuppression following transplantation. Reactivation of latent viruses such as cytomegalovirus (CMV), Epstein-Barr virus (EBV), and Human Herpesvirus 6B (HHV6) are common and often cause symptomatic disease. Reactivations of the polyomaviruses BK virus and JC virus are also common and frequently cause renal disease including hemorrhagic cystitis and less commonly neurologic disease (pervasive multifocal leukoencephalopathy). Respiratory viruses such as adenovirus and human parainfluenza also frequently cause infection. Antiviral pharmacologic agents are only effective against some of these viruses; their use is costly, and associated with significant toxicities and the outgrowth of drug-resistant mutants. As delay in recovery of virus-specific cellular immune response is clearly associated with viral reactivation and disease in these patients, cellular immunotherapy to restore viral-specific immunity is an attractive option that has already been successfully used to target several of these viruses.

To broaden the specificity of single T cells lines to include the three most common viral pathogens of stem cell recipients, the investigators reactivated CMV and adenovirus-specific T cells by using mononuclear cells transduced with a recombinant adenoviral vector encoding the CMV antigen pp65 (Ad5f35CMVpp65). Subsequent stimulations with EBV-LCL transduced with the same vector both reactivated EBV-specific T cells and maintained the expansion of the activated adenovirus and CMV-specific T cells. This method reliably produced T cells with cytotoxic function specific for all three viruses, which the investigators infused into 14 stem cell recipients in a Phase I prophylaxis study. The investigators observed recovery of immunity to CMV and EBV in all patients but an increase in adenovirus-specific T cells was only seen in patients who had evidence of adenovirus infection pre-infusion. A follow-up study in which the frequency of adenovirus-specific T cells was increased in the infused T cells produced similar results, thus highlighting the importance of endogenous antigen to promote the expansion of infused T cells in vivo. Nevertheless, all patients in both clinical trials with pre-infusion CMV, adenovirus or EBV infection or reactivation were able to clear the infection, including one patient with severe adenoviral pneumonia requiring ventilatory support. T cells recognizing multiple antigens can therefore produce clinically relevant effects against all three viruses.

Recent studies have extended the number of targeted viruses, and included HHV6B, BK virus, and Varicella-zoster virus (VZV). In a recent study, 11 patients were treated with VST targeting 5-viruses (CMV, EBV, Adv, HHV6B, BKV) which were generated using a rapid protocol with overlapping peptides encompassing 12 viral protein. VST infusion resulted in a 94% antiviral response rate in these patients (complete or partial responses against CMV=3/3, EBV=5/5, Adv=1/1, HHV6B=2/2, BKV=6/7). Two of the patients who received 5-virus VST developed transplant-associated microangiopathy, which was deemed secondary to HSCT and unrelated to VST infusion. One of these patients developed grade II skin GVHD, which improved with topical therapy. In another recent study, ten adult patients were prophylactically treated with VST specific for CMV, EBV, Adv, and Varicella (VZV). These VSTs were generated using donor-derived dendritic cells which were infected with either Ad5f35-pp65 or with varivax vaccine, and were then pooled and used to stimulate donor PBMCs. All ten patients were protected against EBV, Adv, and VZV. Six patients developed CMV reactivation, but only one required antiviral therapy. Of these 10 patients, 7 developed acute or chronic GVHD, though compared to a non-treated group at the same institution, the rate of GVHD did not differ significantly. Thus, it has been possible to target an extended panel of viruses with a single VST product.

ELIGIBILITY:
Recipient Inclusion Criteria at the Time of Initial VST Infusion and Subsequent Infusions:

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells no earlier than 5 days prior to the date of VST infusion. VSTs administered as:

   1. Prophylaxis for patients at risk of EBV, CMV, adenovirus, HHV6, BKV, JCV and/or HPIV3.
   2. Treatment of reactivation or active infection(s) with EBV, CMV, adenovirus, HHV6, BKV, JCV, and/or HPIV3 that has failed to resolve with at least 14 days of standard antiviral therapy (if available and tolerated). Patients with multiple infections due to the targeted viruses are also eligible.
2. Clinical status at infusion allows for tapering of steroids to less than 0.5 mg/kg/day prednisone or equivalent. 3) Karnofsky/Lansky score of ≥ 50.

4) Bilirubin ≤ 2x, AST ≤5x, Serum creatinine ≤2x upper limit of normal, Hgb ≥8.0 g/dL (level can be achieved with transfusion).

5) Pulse oximetry of > 90% on room air. 6) Available multivirus-specific cytotoxic T lymphocytes 7) Negative pregnancy test (if female of childbearing potential). 8) Patient or parent/guardian capable of providing informed consent.

Recipient Exclusion Criteria at the Time of Initial VST Infusion and Subsequent Infusions

1. Patients with other uncontrolled infections.
2. Patients who received ATG, Campath, Basiliximab or other T cell immunosuppressive monoclonal antibodies within 28 days prior to VST infusion.
3. Received donor lymphocyte infusion or other cellular therapies (with the exception of allogeneic cells related to transplantation) within 28 days prior to VST infusion.
4. Evidence of acute GVHD grades II-IV.
5. Active and uncontrolled relapse of malignancy.
6. Patients with Grade ≥ 3 hyperbilirubinemia.
7. Patients who have received investigational (IND) product within 28 days prior VST infusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute GvHD (grade III-IV) | Within 45 days of the last VSTs dose
  Number of patients with acute GvHD grades III-IV within 45 days of the last dose of VSTs
Incidence of adverse events as per CTCAE common criteria guidelines. | Within 45 days of the last VSTs dose
  2) Grades 3-5 infusion-related adverse events within 45 days of the last dose of VSTs, or 3) Grades 4-5 non-hematological adverse events within 45 days of the last VSTs dose based on a standardized clinical assessment form.

SECONDARY OUTCOMES:
Antiviral response | 1 year
  Peripheral blood and, where relevant, stool and urine will be monitored for viral load by PCR assay. The response in viral load will be defined as follows:
  Complete response: Clearance of targeted virus by PCR assay. Partial response: Decrease in viral load of >= 1 log from baseline Mixed response: Decrease in viral load of >= 1 logarithm from baseline for one targeted infection and an increase or no change in viral load for a second infection.
  Stable disease: Changes insufficient to qualify as partial response or progression Progression: Increase in viral load in body fluids of >= 1 log from baseline or dissemination to other sites of disease.
Antiviral Immunity | 1 year
  Reconstitution of Antiviral Immunity:
  Patient peripheral blood mononuclear cells will be assessed for the presence of virus-reactive T cells using ELIspot and flow cytometry using the MACS Gamma capture kit to assess the percentage of peripheral blood T-cells specific for the targeted virus(es).

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Keller, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Harris KM, Horn SE, Grant ML, Lang H, Sani G, Jensen-Wachspress MA, Kankate VV, Datar A, Lazarski CA, Bollard CM, Keller MD. T-Cell Therapeutics Targeting Human Parainfluenza Virus 3 Are Broadly Epitope Specific and Are Cross Reactive With Human Parainfluenza Virus 1. Front Immunol. 2020 Oct 5;11:575977. doi: 10.3389/fimmu.2020.575977. eCollection 2020. PMID 33123159